CLINICAL TRIAL: NCT06748027
Title: International Expert Consens on Long-term Medical Fasting
Brief Title: Guidelines on Long-term Medical Fasting
Status: Enrolling by invitation | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Software AG Stiftung (Unknown); Reformhaus Stiftung (Unknown); Eden Stiftung (Unknown)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: FastingGuidelines
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-09

CONDITIONS: Fasting Period; Fasting
Keywords: consensus process; long-term fasting
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Fasting — Long-term fasting (>3d)

SUMMARY:
This study will summarize existing clinical practices in long-term medical fasting and provide international expert consensus on their scientific viability

DETAILED DESCRIPTION:
In order to proceed in the most structured and efficient way possible, this project is divided into 6 phases. In the first phase, we intend to use an anonymous survey of international experts in clinical fasting to find out which and how the various fasting methods currently used in clinics and individual clinicians are adapted to the different needs and illnesses of patients. For this purpose, a questionnaire will be drawn up in consultation with individual clinical experts, which will cover the aspects of the various medical fasting therapies in their preparation, implementation and follow-up for a wide range of indications in as much detail as possible. The aim is to cover not only classic therapeutic fasting / fasting according to Otto Buchinger in German-speaking countries, but also fasting therapies as practiced in other European countries, Asia, the USA and Canada. The completed questionnaire will then be filled out anonymously by selected clinics and clinicians.

The findings obtained from the clinical questionnaire will be prepared by the Scientific Committee of the study so that they can be analyzed, evaluated and discussed by international scientists in the field of fasting therapy in the 2nd project phase (two online questionnaire rounds) and 4th project phase (one online questionnaire round and one live discussion) as part of a consensus procedure, more precisely a modified Delphi study. Specific fasting practices that have not yet or not sufficiently been scientifically investigated should also be specifically addressed as part of this project. Their effectiveness is to be studied as quickly as possible in order to be able to carry out fasting therapies in clinics worldwide even more efficiently, safely and simply and to increase the evidence for these integrative medical methods. After initial findings have been obtained in the 2nd project phase through 2 rounds of online questionnaires in the scientific community, a 6-week public consultation phase will follow in which the ( professional) public will comment on the findings obtained up to that point. The results of this external review will be incorporated into the 4th project phase.

After completion of the 3rd and final online questionnaire round, a live discussion will take place among the scientific experts in order to resolve any final discrepancies. Following the evaluation of the live discussion, the Scientific Committee will internally discuss all outstanding points that have arisen from this phase and, if necessary, coordinate any necessary suggestions for changes with all participating experts via email (5th project phase). The final results will then be presented to the public in the form of updated guidelines on medical fasting therapy at a specialist event in summer 2026 and published in a specialist journal (6th project phase).

ELIGIBILITY:
* INCLUSION CRITERIA:

Clinic criteria

* Long-term fasting (≥ 4 days, max. kcal: 25% of daily energy needs*) is offered under medical supervision by medical doctors (MDs) / naturopathic doctors (NDs)
* Long-term fasting has been implemented as a therapeutic intervention for more than 4 years
* ≥ 50 patients / year and / or more than 200 cases in the last 10 years treated with long-term fasting

Personal criteria

* I am a medical doctor (MD) / naturopathic doctor (ND)
* I have 4 years of experience or more in the treatment of patients with long-term fasting (≥ 4 days, max. kcal: 25% of daily energy needs*)
* ≥ 50 patients / year and / or more than 200 cases in the last 10 years treated with long-term fasting

  * according to the recently published fasting terminology in Cell Met.: International consensus on fasting terminology

FASTING REGIMEN DEFINITIONS

· Therapeutic / medically supervised fasting: Therapeutic fasting refers to any fasting regimen that is applied as a therapeutic intervention.

Comment: therapeutic fasting interventions are individually tailored to a person's age, sex, body composition, physical activity level, occupation, goal, and planned duration of fasting.

Medically supervised fasting refers to any fasting regimen that is applied as a therapeutic intervention by a trained physician or similar credentialed healthcare provider.

* Long-term fasting: Prolonged fasting (PF), also called long-term fasting (LTF), refers to fasting regimens lasting ≥4 consecutive days.
* Buchinger therapeutic fasting: Buchinger therapeutic fasting is a fluid-only fasting regimen, allowing for a maximum of 500 kcal/day and lasting at least 5 days, practiced for the prevention or treatment of diseases as well as to support one's individual health, taking into account a person's medical, psychosocial, and spiritual dimensions. It is usually accompanied by bowel/colon cleansing procedures and preceded and followed by a few days of a calorie-restricted, easily digestible diet.
* Fasting-mimicking diet: A fasting-mimicking diet (FMD) specifies any diet specifically composed to induce the metabolic effects of fasting while allowing for a potentially higher caloric intake, including solid foods. It usually refers to a plant-based, calorie-restricted diet with a maximum of approximately 1,000 kcal/day that lasts 3-7 days. FMDs are usually relatively low in refined sugars and starch, low in protein, and high in plant-based fats.
* FX Mayr therapy: FX Mayr therapy or FX-Mayr cure refers to a regimen containing elements of water-only fasting, a very low-calorie diet with a training of "proper chewing" in order to help individuals (re-)gain their sense of satiety, and an easily digestible diet toward the end of the treatment. The dietary intervention is accompanied by bowel cleansing procedures and manual treatments focusing on the abdominal region.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Promising scientific studies on various fasting therapies suggest that fasting will play an important role as a therapeutic method in integrative and complementary medicine in the coming years. To date, however, there are no standardized guidelines for medical fasting therapy. The project presented here aims to address this situation. The aim is to bring together international clinical and scientific experts in the field of fasting in order to develop guidelines for medical fasting as part of a modified Delphi study. The methodology used to develop these guidelines is based on the processes for guidelines defined in the regulations of the Association of Scientific Medical Societies in Germany (AWMF). This project is therefore intended as a basis for the further dissemination and consolidation of this promising integrative medical method.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Consensus on fasting practices | 18 months
  International scientific consensus on clincal fasting practices in long-term medical fasting

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Will try to publish all data in supplements, if journal accepts